CLINICAL TRIAL: NCT06777888
Title: Childhood Obesity Management Using Innovative Digital Technology
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20-00759; PJT - 169013 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2024-12-02; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Obesity Prevention; Child Behaviour; Health Behaviour Change; Obesity and Overweight; Physical Activity
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Healthy Living Program Intervention Group (Experimental)
  Interventions: Behavioral: Family Healthy Living Program weekly group sessions
- Self-Guided Web Only Group (Other)
  Interventions: Behavioral: Self-guided Web Portal Resources Only

INTERVENTIONS:
Behavioral: Family Healthy Living Program weekly group sessions — Children aged 8-12 and at least one caregiver will meet for 9 weekly virtual group intervention sessions (2 hours per session) with program facilitators and will also have access to a virtual Q and A session and up to 3 virtual cooking classes with a Registered Dietician. During the intervention, participants will also have access to digital educational content that is supplementary to what is provided during the individual sessions.
  Other Names: Family Healthy Living Intervention; Early Intervention Program; Generation Health Community
  Arms: Family Healthy Living Program Intervention Group
Behavioral: Self-guided Web Portal Resources Only — Children aged 8-12 and at least one caregiver will be offered access to digital educational content and downloadable resources on topics such as physical activity, healthy eating, and positive mental well-being.
  Arms: Self-Guided Web Only Group

SUMMARY:
The project will evaluate the short- and long-term effects of a 10-week Family Healthy Living Program (FHLP). The program is designed for families with children ages 8-12 years old who are at risk for being above a healthy weight and who would like support with healthy living habits such as physical activity and healthy eating.

Families will participate together, with both parents and children being involved in the program. FHLP participants will receive 9 weekly 2-hour online group sessions with a facilitation team as well as additional web-based resources. They will be compared to a control group of participating families who will be offered only the self-guided web-based resources. This will help us see the impact of offering facilitated FHLP group sessions versus only offering resources online. The FHLP is 10 weeks long, but participants will be followed for 12 months in total so that researchers can look at the long-term impact of participation.

All participating families from both groups will be asked to complete surveys and provide child height and weight measurements at four timepoints: before beginning the program, immediately after completing the program, at 6-months post-program, and at 12-months post-program. Children will also be given FitBit activity watches to measure their daily step counts at each timepoint.

Researchers will compare survey responses, child growth patterns, and FitBit step counts between the FHLP participants and the control group to see whether participating in the FHLP helps families improve their healthy living habits more than only offering a similar curriculum of healthy living resources online for families to access on their own.

ELIGIBILITY:
Inclusion Criteria:

* Children must be aged 8-12 years with at least one primary caregiver who agrees to participate with them. More than one child per parent will be able to participate if the child meets the inclusion criteria.
* Children must have a BMI ≥ 85th percentile for age and sex.

Exclusion Criteria:

* Children below the 85th percentile BMI.
* The inability to communicate (speak, read, and write) in English.
* Any conditions that prevent children from being physically active.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Child BMI Z-scores | From enrollment to 12 month follow-up
  Participants will be asked to self-report measurements of each child's height, weight and age to calculate BMI. Children's BMI z-scores will be calculated based on the World Health Organization criteria. This data will be collected at baseline, 10-week, 6-month and 12-month assessments.

SECONDARY OUTCOMES:
Improving lifestyle behaviours and quality of life in children | From enrollment to 12 month follow-up
  Parents will complete a questionnaire assessing parent support for healthy family lifestyle environment and changes in their child's health-related quality of life. Children will complete questionnaires to assess their physical activity behaviours and dietary behaviours. These questionnaires will be completed at baseline, 10-week, 6-month and 12-month assessments.
Child physical activity measurements | From enrollment to 12 month follow-up
  Changes in physical activity for the child will be measured using FitBit activity trackers. One week of daily step counts will be captured at baseline, 10-week, 6-month and 12-month assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Liu, Principal Investigator — University of Victoria
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be shared with co-investigators.

REFERENCES:
- [Derived] Jantzen RR, Naylor PJ, Strange K, Ball GDC, Masse LC, Rhodes RE, Zhang X, Nolan RP, Zheng S, Rac V, Liu S. Evaluating the Effectiveness of a Family-Based Lifestyle Intervention for Managing Childhood Overweight: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 14;14:e76837. doi: 10.2196/76837. PMID 41085996